CLINICAL TRIAL: NCT04349345
Title: Seminal Fluid's Changes Over Time: a Single Center 20 Years Experience
Brief Title: Seminal Fluid's Changes Over 20 Years
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-01

CONDITIONS: Oligospermia
MeSH Terms: conditions — Oligospermia | interventions — Sperm Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sperm count over time: observation
  Interventions: Diagnostic Test: sperm count

INTERVENTIONS:
Diagnostic Test: sperm count — total progressive sperm motile count

SUMMARY:
This is a cohort study including all the first seminal exams performed at the Fertility Center, Humanitas Research Hospital (Rozzano, Milan) between January 1998 and December 2018.

DETAILED DESCRIPTION:
The objective of this study is to evaluate retrospectively different changes of TPMSC during last 20 years in male population who underwent a seminal exam in our Center

ELIGIBILITY:
Inclusion Criteria:

* male over 18 years old

Exclusion Criteria:

* error in birth or exam date or age under 18,
* abstinence days < 3 or > 6, volume missing o > 10 ml,
* spermatozoa number/ ml missing o >220 x106,
* normal forms missing,
* progressive motility missing

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Male population who underwent a seminal exam in a tertial fertility care center
Sampling Method: Probability Sample
Enrollment: 24395 (Actual)
Dates: Start 1999-01-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Mesaurement of changes of sperm count over time | 20 years
  The objective of this study is to evaluate retrospectively different changes of TPMSC during last 20 years in male population who underwent a seminal exam in a tertial fertility care center, regardless of infertility diagnosis.